CLINICAL TRIAL: NCT04551781
Title: Short Term Low Dose Corticosteroids for Management of Post Covid-19 Pulmonary Fibrosis
Brief Title: Short Term Low Dose Corticosteroids for Management of Post covid19 Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Alaa Rashad, assistant professor of chest diseases and tuberculosis, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVU-MED-CHT019420861
Record Dates: First submitted 2020-09-13; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: Covid-19; post covid-19 fibrosis; low dos steroids
MeSH Terms: conditions — COVID-19 | interventions — Prednisone; Steroids

STUDY DESIGN:
Intervention Model Description: single-blinded randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steroid (Experimental): 20 mg prednisolone for 14 days
  Interventions: Drug: 20 Mg Prednisone for 14 days
- control (Placebo Comparator): controll
  Interventions: Drug: control

INTERVENTIONS:
Drug: 20 Mg Prednisone for 14 days — 20 Mg Prednisone for 14 days
  Other Names: steroid
  Arms: steroid
Drug: control — symptomatic ttt
  Other Names: symptomatic ttt
  Arms: control

SUMMARY:
A randomized controlled trial to study the efficacy of low dose steroid for 14 days in the treatment of post-covid-19 lung infiltrates

DETAILED DESCRIPTION:
: the study included patients with COVID-19 diagnosis with a positive nasopharyngeal swab, they were discharged from quarantine hospitals after 2 Polymerase chain reaction (PCR) swab negative for COVID-19, and have persistent radiological changes in follow-up chest computed tomography (CT) chest, patients with normal CT chest at discharge, patients on chemotherapy, patients <18years old, patients with known interstitial lung disease and patients with rheumatoid arthritis or systemic lupus erythematosus were excluded from the study.

Study patients were randomly assigned to either steroid group or control group and were followed up for 14 days, and CT chest was done at end of 14 days and was evaluated by a radiologist how was blinded for study arm, Ct chest was graded either very minimal infiltrates including reticular shadows, hallow sign, and ground glass s (GGO), infiltrates <25%, and infiltrates >25%.

The steroid group received 20 mg/day prednisolone for 14 days in addition to symptomatic treatment; the control group received symptomatic treatment without steroids Data collected included patient demographics, symptoms, and its duration at baseline, CBC, Ferritin and D-dime, CT chest at discharge, and after 14 days of inclusions in the study.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnosis with a positive nasopharyngeal swab, they were discharged from quarantine hospitals after 2 Polymerase chain reaction (PCR) swab negative for COVID-19, and have persistent radiological changes in follow-up chest computed tomography (CT) chest

Exclusion Criteria:

* patients with normal CT chest at discharge, patients on chemotherapy, patients <18years old, patients with known interstitial lung disease, and patients with rheumatoid arthritis or systemic lupus erythematosus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
improved | 14 days
  resolution of CT chest infiltrates as evaluated by radiologest on a score of no infiltrates, <5%, 5-25%and >25 % infiltrates

CONTACTS AND LOCATIONS:
Overall Officials: alaa DR Rashad, MD, Principal Investigator — south-Vally Universty
Locations (1):
- south-Vally University faculty of medicine, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided